CLINICAL TRIAL: NCT02646852
Title: A Phase I Study of PLX038 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ProLynx LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D15-11073
Record Dates: First submitted 2015-12-31; First posted 2016-01-06 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2019-01

CONDITIONS: Tumors; Neoplasms; Cancer
MeSH Terms: conditions — Neoplasms

ARMS (2):
- PLX038 Q3W (Experimental): intravenous infusion once every 3 weeks
  Interventions: Drug: PLX038
- PLX038 QW ×2 (Experimental): intravenous infusion once weekly for 2 consecutive weeks of a 4-week cycle
  Interventions: Drug: PLX038

INTERVENTIONS:
Drug: PLX038

SUMMARY:
This is a Phase I, open-label, two-arm, dose escalation study of PLX038 intravenous infusion administered to patients with refractory or relapsed solid tumors. This study will explore two different dosing schedules: Arm 1, once every 3 week (q3w), and Arm 2, once weekly for 2 consecutive weeks of a 4-week cycle.

DETAILED DESCRIPTION:
PLX038 is an investigational drug product that has demonstrated reasonable antitumor activity in preclinical colorectal, gastric and lung tumor models in animals. This is a first in human trial to determine the maximum, safest dose of PLX038 IV that can be administered to patients either once every 3 weeks or once every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically (or cytologically)-confirmed diagnosis of solid tumor, refractory after standard therapy for the disease or for which conventional systemic therapy is not reliably effective or no effective therapy is available.
* Aged ≥ 18 years.
* ECOG Performance Status of 0 or 1.
* Adequate clinical laboratory values defined as:

  * absolute neutrophil count ≥ 1.5 × 10^9/L
  * platelets ≥ 100 × 10^9/L
  * hemoglobin ≥ 9.0 g/dL (transfusions permissible)
  * plasma creatinine ≤ 1.5 × upper limit of normal (ULN) for the institution or calculated clearance ≥ 60 mL/min (Cockcroft-Gault formula)
  * bilirubin ≤ 1.5 × ULN
  * alanine transaminase (ALT) and aspartate transaminase (AST) < 2.5 × ULN (< 5 x ULN if documented hepatic metastases)
  * Serum sodium, potassium, magnesium and calcium within normal limits for the institution (supplements may be given to correct values)
* Absence of uncontrolled intercurrent illnesses, including uncontrolled infections, cardiac conditions, or other organ dysfunctions.
* Patients may have measurable or non-measurable disease as defined by RECIST 1.1.
* Signed informed consent prior to the start of any study specific procedures.
* Women of child-bearing potential must have a negative serum or urine pregnancy test. Male and female patients must agree to use acceptable contraceptive methods for the duration of the study and for at least one month after the last drug administration.

Exclusion Criteria:

* Patients will be excluded if they have received previous chemotherapy, immunotherapy, radiotherapy or any other investigational therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) or 5 half-lives for targeted therapies prior to this study entry.
* Have not recovered from adverse events (must be grade ≤1) due to agents administered more than 4 weeks earlier.
* Known hypersensitivity to any study drug component.
* Extensive prior radiotherapy, more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation.
* Any concomitant condition that in the opinion of the investigator could compromise the objectives of this study and the patient's compliance.
* Pregnant or lactating individuals.
* Current malignancies of another type, with the exception of adequately treated in situ cervical cancer and basal cell skin cancer or other malignancies with no evidence of disease for 2 years or more.
* Known history of HIV, HBV or HCV infection.
* Documented or known bleeding disorder.
* Requirement for anticoagulation treatment that increases INR or aPTT above the normal range (low dose DVT or line prophylaxis is allowed).
* Clinically evident CNS metastases or leptomeningeal disease not controlled by prior surgery or radiotherapy; history of seizure disorder not controlled by anti-seizure medication at the time of enrollment. Patients with primary CNS malignancies are excluded.
* Patients with a significant cardiovascular disease or condition, including:

  * Myocardial infarction within 6 months of study entry
  * NYHA Class III or IV heart failure
  * Uncontrolled dysrhythmias or poorly controlled angina.
  * History of serious ventricular arrhythmia (VT or VF, ≥ 3 beats in a row) and/or risk factors (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
  * Baseline prolongation of QT/QTc interval (repeated demonstration of QTc ≥ 450 msec for men and 470 msec for women), or LVEF ≤ 40% by MUGA or ECHO.
* History of clinically significant gastrointestinal bleeding, colitis, or gastrointestinal perforation.
* Patients who require treatment with UGT1A1 inhibitors during the period of investigational treatment with DFP-13318.
* Patients with known Gilbert's syndrome or reduced UGT1A1 activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2023-02 (Actual); Study Completion 2023-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability of PLX038 | Continuous starting on day of first dose (Day 1) up to 30 days after last dose
  Toxicity will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 4.03). Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States